CLINICAL TRIAL: NCT01229514
Title: A Comparison of Functional Magnetic Resonance Imaging (fMRI) Findings in Children With and Without a History of Early Exposure to General Anesthetics
Brief Title: Functional Magnetic Resonance Imaging (fMRI) Findings in Children With Early Exposure to General Anesthesia
Status: Completed | Type: Observational
Sponsor: Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Thomas Taghon, Attending Anesthesiologist, Nationwide Children's Hospital
Other Study IDs: IRB07-00456
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-06

CONDITIONS: Exposed to Anesthesia
Keywords: Children; before; the age of 2 years

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Exposure to anesthesia
  Interventions: Other: fMRI
- Normal controls
  Interventions: Other: fMRI

INTERVENTIONS:
Other: fMRI — fMRI and a response inhibition task to examine activation patterns in the prefrontal cortex and caudate nucleus

SUMMARY:
General anesthetic medications have been shown to cause neuronal cell death in the brains of infant rodents. Ethanol and general anesthetics both act on NMDA and GABA receptors,and appear to have similar mechanisms of toxicity in the immature rodent brain. Functional MRI (fMRI) is a technique developed for mapping brain activation and has been utilized to examine how the brains of children with a history of early exposure to ethanol function differently from children without such a history. This study will utilize fMRI to look for specific changes in brain activation patterns in children with a history of early exposure to general anesthesia, as compared to children without such exposure.

ELIGIBILITY:
Inclusion Criteria:

1. Children ages 10-17 years with an history of exposure to general anesthesia for at least one hour in duration during the ages of 0-24 months of age.
2. The cognitive ability to complete fMRI imaging.
3. Consent of the subject's guardians and assent of the subject.
4. Right hand dominance.
5. English language speaker.

Exclusion Criteria:

1. Subjects with known possibility or knowledge of pregnancy.
2. Documentation of hemodynamic or respiratory instability documented on the anesthetic record
3. Subjects with the inability to complete MRI imaging without sedation.
4. History of prenatal ethanol exposure.
5. History of exposure to antiepileptic medication.
6. History of Attention Deficit Disorder (ADD), or Attention Deficit Hyperactivity Disorder (ADHD)
7. History of traumatic brain injury
8. History of psychiatric disease or exposure to psychoactive medications.
9. History of substance abuse.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from Nationwide Children's Hospital
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Use of fMRI as a tool | one time 10 to 17 yrs. post-anesthesia
  To evaluate the use of fMRI as a tool to investigate the functional consequence of exposure to general anesthetic medications during early brain development

SECONDARY OUTCOMES:
Brain activation patterns | one time 10 to 17 yrs. post-anesthesia
  To compare brain activation patterns in children with and without a history of early exposure to general anesthetic medications while peforming a specific task (go/no-go).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Taghon, DO, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Background] Jevtovic-Todorovic V, Hartman RE, Izumi Y, Benshoff ND, Dikranian K, Zorumski CF, Olney JW, Wozniak DF. Early exposure to common anesthetic agents causes widespread neurodegeneration in the developing rat brain and persistent learning deficits. J Neurosci. 2003 Feb 1;23(3):876-82. doi: 10.1523/JNEUROSCI.23-03-00876.2003. PMID 12574416
- [Background] Mellon RD, Simone AF, Rappaport BA. Use of anesthetic agents in neonates and young children. Anesth Analg. 2007 Mar;104(3):509-20. doi: 10.1213/01.ane.0000255729.96438.b0. PMID 17312200